CLINICAL TRIAL: NCT00948272
Title: Immunogenicity of the Purified Vero Rabies Vaccine - Serum Free in Comparison With the Reference Purified Vero Rabies Vaccine in Pre-exposure Use in Healthy Adults
Brief Title: Study of Purified Vero Rabies Vaccine Serum Free Compared With Reference Purified Vero Rabies Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VRV01; UTN: U1111-1111-4382
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Rabies
Keywords: Rabies; Rabies virus; Purified Vero Rabies Vaccine; Serum Free
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRVg Group (Experimental)
  Interventions: Biological: Purified Vero Rabies Vaccine - Serum Free
- Verorab Group (Active Comparator)
  Interventions: Biological: Purified inactivated rabies vaccine

INTERVENTIONS:
Biological: Purified Vero Rabies Vaccine - Serum Free — 0.5 mL, Intramuscular
  Other Names: VRVg
  Arms: VRVg Group
Biological: Purified inactivated rabies vaccine — 0.5 mL, Intramuscular
  Other Names: Verorab
  Arms: Verorab Group

SUMMARY:
The purpose of this study is to generate data in human on immunogenicity and safety of Purified Vero Rabies Vaccine (VRVg) in support of the vaccine registration.

Primary Objective:

* To demonstrate that VRVg is at least as immunogenic as the reference vaccine, Verorab, in terms of seroconversion rate at Day 42 of the primary vaccination series.

Secondary Objectives:

* To assess the clinical safety of VRVg after each vaccination when administered in a pre-exposure vaccination schedule with a booster at 12 months after the first vaccination in all subjects.
* To describe the immune response induced by VRVg 21 days after two vaccinations in a subset of randomized subjects and 14 days after the last vaccination of the primary vaccination series.

DETAILED DESCRIPTION:
All subjects will receive three vaccinations for primary series and a booster vaccination at 12 months after the first vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 60 years on the day of inclusion
* Provision of a signed Informed Consent Form
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence for at least 4 weeks prior to each vaccination, until at least 4 weeks after each vaccination)
* Entitlement to national social security

Exclusion Criteria :

* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Known human immunodeficiency virus (HIV), Hepatitis B surface (HBs) antigen, or Hepatitis C seropositivity
* Previous vaccination against rabies with any vaccine (in pre- or post-exposure regimen)
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular (IM) vaccination
* Subject at high risk for rabies exposure during the trial period
* Subjects deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment.
* Study site employee who is involved in the protocol and may have direct access to trial related data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of Purified Vero Rabies Vaccine. | 42 days post-primary series vaccination

SECONDARY OUTCOMES:
To provide information concerning the safety after Purified Vero Rabies Vaccine. | 0 to 7 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (6):
- France (6):
  - Gières
  - Montpellier
  - Pierre-Bénite
  - Poitiers
  - Rennes
  - Rueil-Malmaison

REFERENCES:
- [Result] Pichon S, Guinet-Morlot F, Minutello M, Donazzolo Y, Rouzier R, Chassard D, Fitoussi S, Hou V. A serum-free, purified vero cell rabies vaccine is safe and as immunogenic as the reference vaccine Verorab for pre-exposure use in healthy adults: results from a randomized controlled phase-II trial. Vaccine. 2013 Apr 26;31(18):2295-301. doi: 10.1016/j.vaccine.2013.02.058. Epub 2013 Mar 16. PMID 23510665
- See also: Related Info — http://www.sanofipasteur.com